CLINICAL TRIAL: NCT03525587
Title: Development and Validation of a Novel Self-assessment System Based on a Mobile App to Manage Adult Growth Hormone Deficiency (MAGHD App): a Single-Centre Model. GrASS (Growth Hormone Deficiency in Adults Self-assessment System)
Brief Title: Development and Validation of a Self-assessment System Based on a Mobile App to Manage Adult Growth Hormone Deficiency
Acronym: GrASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Vincenzo Rochira, MD, PhD - Associate Professor of Endocrinology, Azienda Ospedaliero-Universitaria di Modena
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 346/17
Record Dates: First submitted 2018-04-17; First posted 2018-05-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Growth Hormone Deficiency
Keywords: Quality Improvement; Quality of Life; Smartphone APP
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Intervention Model Description: Patients with a previous documented AGHD fitting the inclusion/exclusion criteria will be enrolled and grouped as follows:
  * Group 1: patients on long-term r-hGH therapy;
  * Group 2: patients previously treated with r-hGH, who had stopped the treatment for any reason (age, concomitant adverse reactions, contraindications or personal will);
  * Group 3: patients never treated for any reason (according to age, contraindications or lack of patient's consent).
  The whole cohort of AGHD patients (n=100) will undergo 2 consecutive phases: in the first phase (12 months) patients will be evaluated as usual every six months according to our standard clinical practice without using the App and the wearable device (baseline visit, visit 1 and visit 2), while in the second phase (following 12 months) they will be evaluated every six months during the use of the App (visit 3 and visit 4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ongoing r-hGH therapy (Active Comparator): Patients on long-term r-hGH therapy.
  Intervention: Use of "MAGHD App/MAGHD Framework"
  Interventions: Other: Use of "MAGHD App/MAGHD Framework"
- Previous r-hGH therapy (Active Comparator): Patients previously treated with r-hGH, who had stopped the treatment for any reason (age, concomitant adverse reactions, contraindications or personal will).
  Intervention: Use of "MAGHD App/MAGHD Framework"
  Interventions: Other: Use of "MAGHD App/MAGHD Framework"
- Never treated (Active Comparator): Patients never treated for any reason (according to age, contraindications or lack of patient's consent).
  Intervention: Use of "MAGHD App/MAGHD Framework"
  Interventions: Other: Use of "MAGHD App/MAGHD Framework"

INTERVENTIONS:
Other: Use of "MAGHD App/MAGHD Framework" — Patients daily related outcomes will be recorded thanks to the development, implementation and validation of a Smartphone app (MAGHD App) integrated with a software framework able to merge patient's daily activities data on well-being status, QoL, physical activities and sexual function with clinical data collected in their record chart (extrapolated from already available Institutional Databases).

SUMMARY:
Adult Growth Hormone Deficiency (AGHD) is a recognized clinical entity but several barriers concerning patient-clinician communication, inadequate patients' awareness of the disease, low perceived benefit of replacement therapy and poor compliance still remains.

The overall goal of the study is to improve AGHD management through a Smartphone app (MAGHD App: Manage Adult Growth Hormone Deficiency) integrated with a software framework able to merge patients daily data on physical activity, quality of life (QoL), and well-being with clinical data collected in institutional databases. The target population consists of 100 patients with a previous diagnosis of AGHD, whether in treatment with growth hormone or not.

In a prospective 24 months study, MAGHD App will be developed and connected to MAGHD Framework. This system will allow to integrate: 1) Physical Activity Data collected by wearable devices, 2) Patient Related Outcomes Data, periodically inserted by the patients through MAGHD App in response to questions extrapolated from validated questionnaires, 3) HCP Data registered in clinical databases and including medical history, biochemical and radiological examination. Data will converge in MAGHD Framework where they will be analyzed and used to create reports visible to patients (in MAGHD App) and clinicians (by a monitoring dashboard).

The results are expected to positively influence AGHD management by involving patients in care process and giving clinicians a useful tool for clinical practice.

DETAILED DESCRIPTION:
AGHD is widely recognized as a specific clinical entity and recombinant human growth hormone (r-hGH) therapy has become a standard practice since 90s thanks to its beneficial effects on body composition, muscle strength, bone mass, cardiovascular risk and patients' exercise capacity and QoL. All the beneficial effects of r-hGH in AGHD patients have been established mainly on selected populations by both few randomized controlled trials (RCTs) and several clinical trials. Real life studies are also available, but they are mainly based on data collected through multicenter sponsored studies such as the Pharmacia & Upjohn International Metabolic Database (KIMS) and the Hypopituitary Control and Complications Study International Advisory Board (HYPOCCS). All these observational studies suffer from missing data in the original databases and/or lack adequate control group (i.e. untreated GHD patients). Well-conducted real life studies have the advantage to provide information on long-term effects of therapies, as well as on safety, adherence and persistence to therapy. Accordingly, in clinical practice it is common to find a disparity between hormonal levels and patients' subjective well-being: some individuals with a full-blown AGHD do not report any symptom and turn out reluctant to start a treatment, while others with slight GHD experience a deterioration in their QoL that deeply improves after GH replacement. This is mainly due to the fact that clinical presentation of AGHD is frequently based on nonspecific symptoms. Similarly, individual differences in responsiveness to r-hGH are common findings in the real life. Moreover, when other hormonal deficits coexist and patients have to face with a polytherapy, it can be difficult both for clinicians and patients to relate symptoms to the sole AGHD and to verify benefits after treatment. Finally, there is a lack of tools assessing patients' physical activity, which is an important factor to consider when evaluating energy levels, exercise performance, and well-being. Thus, a gap still remains in the real life setting concerning how to measure the improvements occurring in r-hGH treated patients and how to make patients and clinicians more aware of these changes. Nowadays, considering the shortage of established predictive factors for the overall therapeutic response, the decision to whether or not continue treatment depends often on the ratio of perceived and expected beneﬁts over cost and risks of treatment, as well as on the persistent motivation of the patient. These aspects involve also physician's attitude and patient's propensity to start r-hGH replacement therapy. Vice versa the lack of information useful to predict patients' individual response to treatment poses some clinical troubles about how to select patients who may beneficiate from r-hGH therapy. Considering that r-hGH treatment is a chronic therapy requiring a daily self-injection, long-term compliance is still a considerable problem in this setting and is influenced by all the above mentioned issues. It is estimated that about 20 to 30% of patients discontinue the treatment, permanently or for extended periods, making therefore an objective evaluation of the therapeutic effects difficult. All these aspects are enhanced by the paucity of tools available to improve patients' education and awareness of AGHD.

The widespread use of Smartphone applications and wearable devices presents an opportunity to overcome these difficulties in the AGHD management. Although several apps exist to monitor chronic endocrinological diseases, no specific app has been tested in AGHD till now.

In a prospective, 24 months, open-label, monocentric study, an interactive smartphone app (MAGHD App) will be developed, connected to an Integrated Framework (MAGHD Framework) and tested by automatic software testing procedures before the real validation on patients. Subsequently it will be validated on an estimated number of 100 AGHD patients; this system will allow to combine patients' information and HCPs clinical outcomes in a single virtual platform and to return easily accessible data to both AGHD patients and clinicians.

The MAGHD App and the integrated MAGHD Framework will be provided by DataRiver, the research and technological Partner of the study, which is a Contract Research Organization certified by AIFA (Italian drug agency) and accredited as a Research Innovation Institution by the Emilia Romagna Region. The MAGHD software framework will allow integrating patient's Physical Activity data (PA-D), constantly collected by wearable devices (which will be rented and given to patients in the second part of the study), with patient related outcomes data (ePRO-D) and HCP data (HCP-D):

* PA-D will be obtained through wearable devices and will guarantee the automatic collection of data regarding patients' daily life activities. PA recorded by the wearable devices will include: physical activity type, daily steps number, daily walking distance, daily calories burned, sleep duration, sleep quality.
* ePRO-D will be collected via the MAGHD App, which will periodically generate a short question extrapolated from the items of validated questionnaires: AGHDA questionnaire and QLS-H questionnaire for QoL, the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) for well-being evaluation, the International Index of Erectile Function Questionnaire (IIEF-15) and the Female Sexual Function Index (FSFI) for sexual function evaluation (in men and women respectively), the International Physical Activity Questionnaire (IPAQ) for physical activity evaluation and the Pittsburgh Sleep Quality Index (PSQI) for sleep quality evaluation. Additional information on sexual function, working environment, hobbies and adherence to r-hGH therapy (the latter only in Group 1) will be collected through a simple series of questions taken from a specific chart.

The App will record the number of the user answers as well as the missing ones and will periodically provide a visual satisfaction analogue scale on the use of MAGHD App usability. Patients will be notified by the MAGHD App to promptly answer the periodic surveys. The daily surveys could expire after a predefined time interval to prevent the participants to complete them retrospectively, reducing the risk for recall bias.

* HCP data will include:

  * Data obtained from patient's record chart or by interview: anagraphic data, medical history information, comorbidities.
  * Data obtained at baseline and at subsequent visits by physical examination, anthropometric parameters, clinical data and symptoms, r-hGH therapy (weekly dose and duration of therapy in months), if ongoing, other hormone replacement treatments (and relative dosage) in case of multiple pituitary deficits.
  * Data obtained at baseline and at subsequent visits by clinical (biochemical and radiological) examinations:
* pituitary hormones serum levels (IGF-1, insulin-like growth factor binding protein 3, adrenocorticotropic hormone, cortisol, 24-hour urinary free cortisol, thyroid-stimulating hormone, free thyroxine, free triiodothyronine, luteinizing hormone, follicle-stimulating hormone, estradiol and progesterone (in females), testosterone and sex hormone-binding globulin (in men), prolactin;
* biochemical values (haemoglobin, haematocrit, erythrocytes, leukocytes, platelets, renal and hepatic function, electrolytes, glycaemia, TC, HDL-C, LDL-C, triglycerides, bone metabolism);
* dual-energy X-ray absorptiometry (DEXA) scan for assessing body composition, bone mineral content and bone mineral density on whole skeleton, at lumbar site and at femoral site.

The hormonal-biochemical data will be collected at each visit, while the DEXA scan will be performed at baseline, at 12 months and at the end of the study.

PA-D, ePRO-D and HCP-D will converge in the MAGHD Framework where they will be integrated, analyzed and used to create graphs and tables visible both to patients (in MAGHD App) and clinicians (by a monitoring dashboard).

Patients will receive periodically a feedback concerning: i) %change of their QoL, well-being, sleep quality, sexual function and ii) changes in daily physical activities. This kind of report will enhance patient's awareness on day-by-day changes related to their clinical condition. In particular frequent feedback on QoL and well-being will provide a more objective evaluation of these parameters, thus minimizing possible interference due to life events occurred close to the day in which the questionnaires are filled. Moreover, a summary of the patient's clinical outcomes will be provided through the MAGHD App in a simple graphical way in order to communicate changes in serum IGF-1 and lipid profile.

The project will be carried out in 24 months. Months 1-6 will focus on: 1) App development, 2) Integrated Framework development, 3) App testing.

Patient enrollment and baseline visits will occur between months 1 and 6, then six-month visits (visit 1, visit 2, visit 3 and visit 4) will occur in the next 2 years. In the first phase (12 months) the recruited patients, after having signed the informed consent, will be followed every six months according to our normal clinical practice without using the App and the wearable device (baseline, visit 1 and visit 2). Then they will be trained to use the MAGHD App prior to enter the second phase (following 12 months), in which they will be evaluated every six months during the use of the App and the wearable device (visit 3 and visit 4).

HCP data will be collected both in phase 1 (usual follow-up without the use of MAGHD App) and phase 2 (during the use of MAGHD App). Anamnestic, clinical and biochemical data will be collected at each visit (baseline, visit 2, visit 3, visit 4), while DEXA scan (radiological data) will be performed only twice (at baseline and at the end of the protocol).

All the other data will be collected differently in the two consecutive phases:

* QoL and well-being data:

  * In Phase 1 AGHDA questionnaire, QLS-H questionnaire and WEMWBS will be administered to patients in paper form at baseline, visit 1 and visit 2.
  * In Phase 2 MAGHD App will periodically generate a short question extrapolated from the items of the same validated questionnaires.
* Sexual function:

  * In Phase 1 IIEF-5 questionnaire (for men) and FSFI questionnaire (for woman) will be administered to patients in paper form at baseline, visit 1 and visit 2.
  * In Phase 2 MAGHD App will periodically generate a short question extrapolated from the items of the same validated questionnaires.
* Physical activity and sleep quality:

  * In Phase 1 physical activity will be evaluated through the IPAQ questionnaire and sleep quality through the PSQI questionnaire; both will be administered to patients in paper form at baseline, visit 1 and visit 2.
  * In Phase 2 MAGHD App will periodically generate a short question extrapolated from the items of the same validated questionnaires; data on physical activity and sleep quality will be also automatically collected through wearable devices.
* Additional information on sexual function, working environment, hobbies and adherence to r-hGH therapy (the latter only in Group 1):

  * In Phase 1 these aspects will be evaluated at baseline, visit 1 and visit 2, through a specific chart in paper form.
  * In Phase 2 the same questions will be sent through the MAGHD App.

ELIGIBILITY:
Inclusion Criteria:

1. Having a documented diagnosis of AGHD, according to the latest Endocrine Society clinical practice guidelines
2. Being at least 18 years old
3. Having a good Italian understanding
4. Owing smartphones with either an Android or iPhone operating system
5. Patients with other pituitary deficits will be enrolled only if the other hormonal deficiencies are well controlled by replacement treatments since six months in order to avoid the overlap of effects due to different therapies.

Exclusion Criteria:

1) Patients who do not plan to continue follow-up at the Endocrinology Unit of Modena 2) Patients with a diagnosis of biochemical GHD outside the appropriate clinical context of pituitary disease 3) Patients with major psychiatric diseases, chronic highly invalidating diseases (these patients will be considered not eligible for being enrolled in the study due to the impact of the underlying disease on well-being and daily activities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of quality of life (QoL) from baseline | 24 months
  Comparison of changes of QoL score from baseline for each patient within the three different groups. QoL score will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.

SECONDARY OUTCOMES:
Changes of well-being from baseline | 24 months
  Comparison of changes of Well-being score from baseline for each patient within the three different groups. Well-being score will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of physical activity from baseline | 24 months
  Comparison of changes of physical activity score from baseline for each patient within the three different groups. Physical activity score will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of sleep quality from baseline | 24 months
  Comparison of changes of sleep quality score from baseline for each patient within the three different groups. Sleep quality score will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of sexual function from baseline | 24 months
  Comparison of changes of sexual function scores (IIEF-5 score for men and FSFI score for woman) from baseline for each patient within the three different groups. Sexual function scores will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of insulin-like growth factor 1 (IGF-1) levels from baseline | 24 months
  Comparison of changes of IGF-1 levels from baseline for each patient within the three different groups. IGF-1 levels will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of lipid profile from baseline | 24 months
  Comparison of changes of total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides from baseline for each patient within the three different groups. Lipid profile will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of body composition from baseline | 24 months
  Comparison of changes of % of lean mass and fat mass from baseline for each patient within the three different groups. Body composition will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Changes of bone mineral density from baseline | 24 months
  Comparison of changes of T-score at lumbar site and at femoral site from baseline for each patient within the three different groups. Bone mineral density will be evaluated and compared before and after the use of the integrated system MAGHD App/MAGHD Framework.
Adherence to r-hGH therapy (average number of weekly forgetfulnesses) | 24 months
  Evaluation of possible changes in adherence to r-hGH therapy (only in patients of Group 1) from Phase 1 and Phase 2.
  Average number of weekly forgetfulnesses of r-hGH therapy will be considered to verify the adherence to therapy.
Impact of physical activity on BMI | 12 months
  Evaluation of the impact of physical activity in AGHD patients (as recorded by the MAGHD App in Phase 2) on BMI. Weight and height will be combined to report BMI in kg/m^2.
Impact of physical activity on body composition | 12 months
  Evaluation of the impact of physical activity in AGHD patients (as recorded by the MAGHD App in Phase 2) on body composition (% of lean mass and fat mass).
Impact of physical activity on lipid profile | 12 months
  Evaluation of the impact of physical activity in AGHD patients (as recorded by the MAGHD App in Phase 2) on lipid profile (total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides).
User's satisfaction about MAGHD App | 12 months
  Evaluation of user's satisfaction about MAGHD App through the number of messages the user has returned in response to the questions of each questionnaire he received. The App will record the number of the user answers as well as the missing ones. For each patient will be considered the following ratio: number of returned messeges/total number of sent messages.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Rochira, Professor, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (1):
- Azienda Ospedaliero - Universitaria di Modena, Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The University of Modena and Reggio Emilia and the P.I. are the owners of the study data, which will be available for DataRiver for the results' analysis. The project will be disseminated through publication on indexed international journals and will be evaluated by number of papers/citations received in scientific and academic context. Preliminary results will be shown at National and International congresses.

REFERENCES:
- [Background] Ho KK; 2007 GH Deficiency Consensus Workshop Participants. Consensus guidelines for the diagnosis and treatment of adults with GH deficiency II: a statement of the GH Research Society in association with the European Society for Pediatric Endocrinology, Lawson Wilkins Society, European Society of Endocrinology, Japan Endocrine Society, and Endocrine Society of Australia. Eur J Endocrinol. 2007 Dec;157(6):695-700. doi: 10.1530/EJE-07-0631. PMID 18057375
- [Background] Molitch ME, Clemmons DR, Malozowski S, Merriam GR, Vance ML; Endocrine Society. Evaluation and treatment of adult growth hormone deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jun;96(6):1587-609. doi: 10.1210/jc.2011-0179. PMID 21602453
- [Background] Woodhouse LJ, Mukherjee A, Shalet SM, Ezzat S. The influence of growth hormone status on physical impairments, functional limitations, and health-related quality of life in adults. Endocr Rev. 2006 May;27(3):287-317. doi: 10.1210/er.2004-0022. Epub 2006 Mar 16. PMID 16543384
- [Background] van Bunderen CC, van Varsseveld NC, Erfurth EM, Ket JC, Drent ML. Efficacy and safety of growth hormone treatment in adults with growth hormone deficiency: a systematic review of studies on morbidity. Clin Endocrinol (Oxf). 2014 Jul;81(1):1-14. doi: 10.1111/cen.12477. Epub 2014 May 12. PMID 24750271
- [Background] Hoybye C, Christiansen JS. Growth hormone replacement in adults - current standards and new perspectives. Best Pract Res Clin Endocrinol Metab. 2015 Jan;29(1):115-23. doi: 10.1016/j.beem.2014.09.006. Epub 2014 Oct 2. PMID 25617177
- [Background] Newman CB, Carmichael JD, Kleinberg DL. Effects of low dose versus high dose human growth hormone on body composition and lipids in adults with GH deficiency: a meta-analysis of placebo-controlled randomized trials. Pituitary. 2015 Jun;18(3):297-305. doi: 10.1007/s11102-014-0571-z. PMID 24810900
- [Background] Bengtsson BA, Abs R, Bennmarker H, Monson JP, Feldt-Rasmussen U, Hernberg-Stahl E, Westberg B, Wilton P, Wuster C. The effects of treatment and the individual responsiveness to growth hormone (GH) replacement therapy in 665 GH-deficient adults. KIMS Study Group and the KIMS International Board. J Clin Endocrinol Metab. 1999 Nov;84(11):3929-35. doi: 10.1210/jcem.84.11.6088. PMID 10566630
- [Background] Attanasio AF, Bates PC, Ho KK, Webb SM, Ross RJ, Strasburger CJ, Bouillon R, Crowe B, Selander K, Valle D, Lamberts SW; Hypoptiuitary Control and Complications Study International Advisory Board. Human growth hormone replacement in adult hypopituitary patients: long-term effects on body composition and lipid status--3-year results from the HypoCCS Database. J Clin Endocrinol Metab. 2002 Apr;87(4):1600-6. doi: 10.1210/jcem.87.4.8429. PMID 11932289
- [Background] Alexopoulou O, Abs R, Maiter D. Treatment of adult growth hormone deficiency: who, why and how? A review. Acta Clin Belg. 2010 Jan-Feb;65(1):13-22. doi: 10.1179/acb.2010.002. PMID 20373593
- [Background] Lazure P, Bartel RC, Biller BM, Molitch ME, Rosenthal SM, Ross JL, Bernsten BD, Hayes SM. Contextualized analysis of a needs assessment using the Theoretical Domains Framework: a case example in endocrinology. BMC Health Serv Res. 2014 Jul 24;14:319. doi: 10.1186/1472-6963-14-319. PMID 25060235
- [Background] Buijink AW, Visser BJ, Marshall L. Medical apps for smartphones: lack of evidence undermines quality and safety. Evid Based Med. 2013 Jun;18(3):90-2. doi: 10.1136/eb-2012-100885. Epub 2012 Aug 25. PMID 22923708
- [Background] Cui M, Wu X, Mao J, Wang X, Nie M. T2DM Self-Management via Smartphone Applications: A Systematic Review and Meta-Analysis. PLoS One. 2016 Nov 18;11(11):e0166718. doi: 10.1371/journal.pone.0166718. eCollection 2016. PMID 27861583
- [Background] Chin SO, Keum C, Woo J, Park J, Choi HJ, Woo JT, Rhee SY. Successful weight reduction and maintenance by using a smartphone application in those with overweight and obesity. Sci Rep. 2016 Nov 7;6:34563. doi: 10.1038/srep34563. PMID 27819345
- [Background] Ryan EA, Holland J, Stroulia E, Bazelli B, Babwik SA, Li H, Senior P, Greiner R. Improved A1C Levels in Type 1 Diabetes with Smartphone App Use. Can J Diabetes. 2017 Feb;41(1):33-40. doi: 10.1016/j.jcjd.2016.06.001. Epub 2016 Aug 25. PMID 27570203
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760